CLINICAL TRIAL: NCT01235572
Title: Phase 2 Study of Early Discharge and Outpatient Management of Adult Patients Following Intensive Chemotherapy for MDS and Non-APL AML
Brief Title: Early Discharge and Outpatients Care in Patients With Myelodysplastic Syndrome or Acute Myeloid Leukemia Previously Treated With Intensive Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2449.00; NCI-2012-03028 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2449.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium)
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2015-02

CONDITIONS: Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia with multilineage dysplasia following myelodysplastic syndrome; Adult acute eosinophilic leukemia; Adult acute basophilic leukemia; De; novo myelodysplastic syndromes; Secondary myelodysplastic syndromes; Untreated adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Basophilic, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Health services research (early discharge, outpatient care) (Experimental): Patients are discharged within 72 hours after completion of chemotherapy and undergo standard outpatient care by a RN, PA, or resident/fellow at a local facility or the study center approximately 3 times per week, as clinically indicated for up to 45 days.
  Interventions: Procedure: standard follow-up care; Other: medical chart review; Procedure: quality-of-life assessment

INTERVENTIONS:
Procedure: standard follow-up care — Undergo early discharge and standard outpatient care
Other: medical chart review — Undergo early discharge and standard outpatient care
  Other Names: chart review
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This phase II trial studies how well early discharge and outpatient care works in patients with myelodysplastic syndrome or acute myeloid leukemia previously treated with intensive chemotherapy. Gathering information about patients with myelodysplastic syndrome or acute myeloid leukemia who are discharged after finishing chemotherapy, or who stay in the hospital until blood counts return to normal, may help doctors learn more about the safety of allowing patients to leave the hospital early, the patient's quality of life, use of medical services, and the cost of these services associated with such a policy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate the early death rate in patients discharged after completion of intensive induction or salvage chemotherapy.

SECONDARY OBJECTIVES:

I. Compare the costs incurred by patients discharged early after induction or salvage chemotherapy with similar patients who are discharged only after their blood counts recover.

II. Compare resource utilization (transfusions, etc.) in patients discharged early after induction or salvage chemotherapy with similar patients who are discharged only after blood count recovery.

III. Compare the quality of life in patients discharged early after induction or salvage chemotherapy with similar patients who are discharged only after their blood counts recover.

OUTLINE:

Patients are discharged within 72 hours after completion of chemotherapy and undergo standard outpatient care by a registered nurse (RN), physician assistant (PA), or resident/fellow at a local facility or the study center approximately 3 times per week, as clinically indicated for up to 45 days.

After completion of study, patients are followed up for 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of myelodysplastic syndromes (MDS) or acute myeloid leukemia (AML) other than acute promyelocytic leukemia (APL) with t(15;17)(q22;q12), (promyelocytic leukemia [PML]/retinoic acid receptor [RAR]), or variants according to the 2008 World Health Organization (WHO) classification
* Currently undergoing AML-like intensive induction or re-induction chemotherapy, or is planned to start such therapy within 1 week
* Provide signed written informed consent
* Patients can be repeatedly enrolled in this protocol (e.g. for induction and 1st or subsequent salvage therapy)

Exclusion Criteria:

* Drug hypersensitivities or allergies disabling use of prophylactic antimicrobials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Proportion of early deaths among patients who are discharged after completion of induction or salvage chemotherapy | Up to day 35
  A one-sided lower exact 95% confidence interval for the proportion of early deaths after discharge will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Roland Walter, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States